CLINICAL TRIAL: NCT00837876
Title: A Phase II Trial of Sorafenib and Erlotinib in Unresectable Pancreatic Cancer
Brief Title: Sorafenib and Erlotinib in Treating Patients With Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jordan Berlin, MD, Professor of Medicine; Clinical Director, GI Oncology Program; Director, Phase I Program; Medical Director, Clinical Trials Shared Resources; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0815; P30CA068485 (NIH); VU-VICC-GI-0815
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2013-07

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Sorafenib + Erlotinib
  Interventions: Drug: Sorafenib; Drug: Erlotinb

INTERVENTIONS:
Drug: Sorafenib — 400 mg taken by mouth 1 time per day.
Drug: Erlotinb — 150 mg taken by mouth 1 time per day.

SUMMARY:
RATIONALE: Sorafenib and erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sorafenib together with erlotinib works in treating patients with pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of sorafenib tosylate in combination with erlotinib hydrochloride in patients with unresectable pancreatic cancer.

Secondary

* To determine the response rate in patients treated with this regimen.
* To determine the progression-free survival of patients treated with this regimen at 4 months.
* To evaluate the safety profile of this regimen in these patients.
* To evaluate the change in serum Ca 19-9 levels at baseline and at 8-week intervals.
* To evaluate the plasma proteomic profile at baseline and at 8 weeks to correlate with clinical parameters in order to identify potential prognostic or predictive markers.
* To analyze single-nucleotide polymorphisms on DNA obtained from pretreatment blood samples to evaluate toxicity and response to erlotinib hydrochloride.

OUTLINE: Patients receive oral sorafenib tosylate once or twice daily and oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Serum samples are collected at baseline and at 8-week intervals to measure Ca 19-9 levels, and plasma and buffy coat samples are collected at baseline and at week 8 for proteomic assessment and genotyping of single-nucleotide polymorphisms associated with response and toxicity to erlotinib hydrochloride.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Microscopically confirmed diagnosis of pancreatic adenocarcinoma

  * Unresectable disease
  * No neuroendocrine tumors or cystadenocarcinoma
* Measurable or evaluable disease by RECIST criteria
* No known brain metastases

  * Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* Creatinine ≤ 1.5 times ULN
* INR < 1.5 or PT/PTT normal unless patients are receiving anticoagulation treatments
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception before, during, and for at least 6 months after completion of study treatment
* Able to swallow whole pills
* No patients who currently smoke
* No cardiac disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New-onset angina (began within the past 3 months)
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension defined as systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal medical management
* No arterial thrombotic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 in the past 4 weeks
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 in the past 4 weeks
* No significant traumatic injury in the past 4 weeks
* No known untreated malabsorption problem (e.g., ulcerative colitis, Crohn's disease)
* No known HIV positivity or chronic hepatitis B or C
* No known or suspected allergy to sorafenib tosylate or erlotinib hydrochloride
* No active clinically serious infection > CTCAE grade 2
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy (except for cancer-related blood clots)
* No dermatitis ≥ CTCAE grade 2 at baseline
* No patients who currently smoke

PRIOR CONCURRENT THERAPY:

* No prior treatment with antiangiogenics (e.g., bevacizumab, thalidomide, marimastat, interferon alfa, vatalanib, vandetanib, ZD6126, sorafenib, semaxanib, sunitinib, axitinib)
* No more than one line of prior therapy for metastatic disease
* More than 4 weeks since prior major surgery or open biopsy
* No concurrent strong CYP34A inhibitors or inducers
* Concurrent warfarin or heparin allowed with the approval of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D. Berlin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Purchase Cancer Group - Paducah, Paducah, Kentucky
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - Baptist Regional Cancer Center at Baptist Riverside, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from October 2008 until February 2011.
Pre-assignment Details: 37 patients consented and went on study. Six patients were ineligible.
Period: Overall Study
Arm/Group | Treatment
Started | 37
Completed | 0
Not Completed | 37
Not completed — Death | 2
Not completed — Adverse Event | 7
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — disease progression | 24

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Progression-free Survival
Description: Number of patients with progression-free survival at 8 weeks
Time Frame: at 8 weeks
Population: Patients who received treatment for >= 8 weeks. 14 study patients were treated for < 8 weeks due to toxicity (5), disease progression (5), did not receive study drug (1), respiratory failure (1), drug held more than 28 days (1), patient withdrawal (1). The remaining 13 participants did not have a progression-free survival at 8 weeks.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 23
participants | 10

2. Secondary Outcome: Response Rate
Description: Per RECIST criteria v. 1.0: measurable lesions: CR disappearance of target lesions, PR > 30% decrease in the sum of the longest diameter (LD) of target lesions, PD > 20% increase in the sum of the LD of target lesions or appearance of new lesions, SD neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: at 4 months
Population: Participants who received treatment for 4 or more months. The remaining 10 participants received treatment for less than 4 months and were not evaluable.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 8
  Progressive Disease | 19

3. Secondary Outcome: Number of Patients With Progression-free Survival
Description: Participants with progression-free survival at 4 months.
Time Frame: at 4 months
Population: Patients with progression-free survival at 4 months. The remaining 17 patients were not available for evaluation at 4 months due to toxicity (5), disease progression (5), patient withdrawal (1),respiratory failure (1), study drug held more than 28 days (1), and no study drug (1.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
participants | 4

4. Secondary Outcome: Number of Patients With Worst Grade Toxicities
Description: Number of patients with worst-grade toxicity at each of five grades (grade 1 to 5, with 5 most severe) following NCI Common Toxicity Criteria: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death.
Time Frame: every 4 weeks and every 8 weeks in follow-up to resolution of toxicity
Population: All patients who received treatment with the study drugs. One patient did not receive treatment.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
participants
  number of patients with worst grade toxicity - 1 | 1
  number of patients with worst grade toxicity - 2 | 5
  number of patients with worst grade toxicity - 3 | 26
  number of patients with worst grade toxicity - 4 | 3
  number of patients with worst grade toxicity - 5 | 1

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 27/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=37)
nausea (Gastrointestinal disorders) | 9 (14)
vomiting (Gastrointestinal disorders) | 7 (11)
acidosis (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 5 (7)
Pain, NOS (General disorders) | 5 (10)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
death - NOS (General disorders) | 2 (2)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
infection with unknown ANC, artery (Infections and infestations) | 1 (1)
bladder infection (Infections and infestations) | 1 (1)
infection, normal ANC (Infections and infestations) | 1 (1)
infection, Hickman catheter (Infections and infestations) | 1 (1)
hyperbilirubinemia (Metabolism and nutrition disorders) | 5 (6)
hemoglobin (Investigations) | 2 (3)
fatigue (General disorders) | 4 (4)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
confusion (Psychiatric disorders) | 5 (7)
calcium, serum-low-hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
pain in abdomen (Gastrointestinal disorders) | 10 (15)
diarrhea (Gastrointestinal disorders) | 2 (2)
enteritis (Gastrointestinal disorders) | 1 (1)
hypocalcemia (Pregnancy, puerperium and perinatal conditions) | 1 (1)
hypochloremia (Metabolism and nutrition disorders) | 1 (1)
thrombosis (Vascular disorders) | 2 (2)
hemorrhage, GI (Gastrointestinal disorders) | 1 (1)
fever (General disorders) | 2 (2)
pain, right upper quadrant (General disorders) | 2 (2)
infection with unknown ANC, blood (Infections and infestations) | 2 (2)
infection with unknown ANC, wound (Infections and infestations) | 1 (1)
AST, SGOT (Metabolism and nutrition disorders) | 2 (2)
alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
obstruction, GI (Gastrointestinal disorders) | 1 (1)
infection with unknown ANC, lung (Infections and infestations) | 1 (2)
cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
pain in back (Musculoskeletal and connective tissue disorders) | 3 (4)
distension, abdominal (Gastrointestinal disorders) | 1 (1)
pulmonary, upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pain in stomach (Gastrointestinal disorders) | 1 (1)
edema, limb (General disorders) | 1 (1)
ammonia level increase (Metabolism and nutrition disorders) | 1 (1)
appendicitis (Infections and infestations) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (N=37)
diarrhea (Gastrointestinal disorders) | 21 (40)
nausea (Gastrointestinal disorders) | 15 (22)
anorexia (Metabolism and nutrition disorders) | 14 (19)
vomiting (Gastrointestinal disorders) | 10 (11)
dehydration (Gastrointestinal disorders) | 9 (11)
mucositis/stomatitis (Gastrointestinal disorders) | 9 (10)
constipation (Gastrointestinal disorders) | 8 (8)
flatulence (Gastrointestinal disorders) | 8 (10)
heartburn/dyspepsia (Gastrointestinal disorders) | 2 (3)
fatigue (General disorders) | 22 (42)
weight loss (Metabolism and nutrition disorders) | 12 (17)
hyperglycemia (Metabolism and nutrition disorders) | 19 (36)
alkaline phosphatase (Investigations) | 18 (25)
AST, SGOT (Metabolism and nutrition disorders) | 14 (27)
ALT, SGPT (Metabolism and nutrition disorders) | 13 (24)
hyponatremia-sodium, low (Metabolism and nutrition disorders) | 10/13 (13)
hypokalemia (Metabolism and nutrition disorders) | 9 (15)
hyperbilirubinemia (Metabolism and nutrition disorders) | 8 (19)
hypocalcemia (Metabolism and nutrition disorders) | 6 (8)
hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 4 (10)
hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
hemoglobin (Investigations) | 17 (33)
lymphopenia (Investigations) | 12 (30)
platelets (Investigations) | 8 (11)
leukocytes (Metabolism and nutrition disorders) | 5 (9)
rash-acne/acneiform (Skin and subcutaneous tissue disorders) | 17 (22)
dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
rash-hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 (18)
pain, abdomen NOS (Gastrointestinal disorders) | 9 (20)
pain, back (Musculoskeletal and connective tissue disorders) | 6 (8)
pain, headaches (Nervous system disorders) | 3 (3)
dysarthria/voice changes (Nervous system disorders) | 6 (7)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
confusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
depression (Psychiatric disorders) | 3 (3)
Neuropathy-sensory (Nervous system disorders) | 3 (4)
edema limb (General disorders) | 3 (3)
constitutional symptoms, other (General disorders) | 7 (21)
albumin, serum-low (Metabolism and nutrition disorders) | 15 (21)
glucose, serum-high-hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
Taste alteration (Gastrointestinal disorders) | 3 (4)
fever (in the absence of neutropenia , where neutropenia is defined as ANC<1.0 x 10e9/L) (Infections and infestations) | 3 (4)
Insomnia (Nervous system disorders) | 2 (2)
sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Metabolic/Laboratory, other (Metabolism and nutrition disorders) | 2 (3)
dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 3 (5)
Pruritis, itching (Skin and subcutaneous tissue disorders) | 2 (2)
Pain-chest/thorax (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pain-sinus (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pain-throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory, other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 6 (10)
Infection-other (Infections and infestations) | 2 (3)
Infection with unknown ANC-upper airway NOS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3 (3)
Vascular-other (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes